CLINICAL TRIAL: NCT00064701
Title: A Phase III, Randomized, Open-Label, Comparative, Multi-Center Study to Assess the Safety and Efficacy of Prograf (Tacrolimus)/MMF, Modified Release (MR) Tacrolimus/MMF and Neoral (Cyclosporine)/MMF in de Novo Kidney Transplant Recipients
Brief Title: Comparative Study of Modified Release (MR) Tacrolimus/Mycophenolate Mofetil (MMF) in de Novo Kidney Transplant Recipients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02-0-158
Record Dates: First submitted 2003-07-10; First posted 2003-07-14 (Estimated); Results first posted 2013-09-26 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-11

CONDITIONS: Kidney Transplantation
Keywords: De Novo Kidney Transplant; cyclosporine; Prograf®; mycophenolate mofetil; tacrolimus
MeSH Terms: interventions — Tacrolimus; Cyclosporine; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tacrolimus (Experimental): Participants received a first dose of tacrolimus between 0.075 and 0.10 mg/kg twice daily, orally prior to or within 48 hours of the completion of the transplant procedure, and subsequently as twice daily oral doses adjusted based on clinical evidence of efficacy, blood concentrations of tacrolimus and adverse events. Participants also received 1.0 g mycophenolate mofetil orally twice daily throughout the study.
  Interventions: Drug: Tacrolimus; Drug: mycophenolate mofetil
- Tacrolimus Modified Release (Active Comparator): Participants received a first dose of tacrolimus modified release between 0.15 and 0.20 mg/kg/day, given as a single oral dose in the morning, prior to or within 48 hours following the completion of the transplant procedure, and subsequently as once daily oral doses adjusted based on clinical evidence of efficacy, blood concentrations of tacrolimus and adverse events. Participants also received 1.0 g mycophenolate mofetil orally twice daily throughout the study.
  Interventions: Drug: Tacrolimus Modified Release (MR); Drug: mycophenolate mofetil
- Cyclosporine (Active Comparator): Participants received a first dose of cyclosporine between 4 to 5 mg/kg orally prior to or within 48 hours following the completion of the transplant procedure and subsequently as twice daily oral doses adjusted based on clinical evidence of efficacy, blood concentrations of tacrolimus and adverse events. Participants also received 1.0 g mycophenolate mofetil orally twice daily throughout the study.
  Interventions: Drug: cyclosporine microemulsion; Drug: mycophenolate mofetil

INTERVENTIONS:
Drug: Tacrolimus Modified Release (MR) — The target range for whole blood tacrolimus trough concentrations was 7 to 16 ng/mL for days 0 through 90, and 5 to 15 ng/mL thereafter.
  Other Names: Advagraf, FK506, FKMR, MR4, Astagraf XL
  Arms: Tacrolimus Modified Release
Drug: Tacrolimus — The target range for whole blood tacrolimus trough concentrations was the recommended trough concentration range for Prograf: 7 to 16 ng/mL for days 0 through 90 and 5 to 15 ng/mL thereafter.
  Other Names: Prograf, FK506
  Arms: Tacrolimus
Drug: cyclosporine microemulsion — The target range for whole blood cyclosporine trough concentrations was 125 to 400 ng/mL for days 0 through 90, and 100 to 300 ng/mL thereafter.
  Other Names: Neoral, CsA
  Arms: Cyclosporine
Drug: mycophenolate mofetil — Oral
  Other Names: CellCept, MMF

SUMMARY:
The purpose of this study is to compare the safety and efficacy of tacrolimus/mycophenolate mofetil (MMF), cyclosporine/MMF and tacrolimus modified release/MMF in de novo kidney transplant recipients.

DETAILED DESCRIPTION:
This was a 3 arm randomized, open-label, comparative, multi-center study in de novo kidney transplant recipients at 60 centers in the U.S., Canada and Brazil.

The study consisted of a 1-year post-transplant efficacy and safety study with a clinical continuation phase of a minimum of 2 years or until commercial availability of tacrolimus modified release, unless the Data Safety Monitoring Board or sponsor specified otherwise.

ELIGIBILITY:
Inclusion Criteria:

* Recipient of a primary or retransplanted non-human leukocyte antigen (HLA)-identical living or non-HLA-identical cadaveric kidney transplant
* Age greater or equal to 12 years

Exclusion Criteria:

* Recipient or donor is known seropositive for human immunodeficiency virus (HIV)
* Has current malignancy or history of malignancy
* Has significant liver disease
* Has uncontrolled concomitant infection or any other unstable medical condition
* Is receiving everolimus or enteric coated mycophenolic acid at any time during the study
* Received kidney with a cold ischemia time of equal or more than 36 hours
* Received kidney transplant from a cadaveric donor equal or more than 60 years of age
* Received intravenous immunoglobulin (IVIG) therapy prior to randomization

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 668 (Actual)
Dates: Start 2003-06; Primary Completion 2005-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Global Development
Locations (46):
- United States (39):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Loma Linda, California
  - Los Angeles, California
  - Palo Alto, California
  - San Diego, California
  - San Francisco, California
  - Denver, Colorado
  - Washington D.C., District of Columbia
  - Gainesville, Florida
  - Jacksonville, Florida
  - Augusta, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Lexington, Kentucky
  - New Orleans, Louisiana
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Livingston, New Jersey
  - New Brunswick, New Jersey
  - Albany, New York
  - Buffalo, New York
  - New York, New York
  - Valhalla, New York
  - Chapel Hill, North Carolina
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Portland, Oregon
  - Harrisburg, Pennsylvania
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Fairfax, Virginia
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Brazil (3):
  - Porto Alegre
  - Rio de Janeiro
  - São Paulo
- Canada (4):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Toronto, Ontario
  - Montreal, Quebec

REFERENCES:
- [Background] Silva HT Jr, Yang HC, Abouljoud M, Kuo PC, Wisemandle K, Bhattacharya P, Dhadda S, Holman J, Fitzsimmons W, First MR. One-year results with extended-release tacrolimus/MMF, tacrolimus/MMF and cyclosporine/MMF in de novo kidney transplant recipients. Am J Transplant. 2007 Mar;7(3):595-608. doi: 10.1111/j.1600-6143.2007.01661.x. Epub 2007 Jan 11. PMID 17217442

RESULTS

PARTICIPANT FLOW:
Recruitment Details: De novo kidney transplant recipients 12 years of age and older were randomized in a 1:1:1 ratio to 1 of 3 treatment arms.
Pre-assignment Details: This study was a 1-year safety and efficacy study followed by a clinical continuation phase that continued until the sponsor discontinued the study in March 2009.
Period: One Year Post-transplant
Arm/Group | Tacrolimus | Tacrolimus Modified Release | Cyclosporine
Started | 219 | 226 | 223
Received Study Drug | 212 | 214 | 212
Completed | 179 | 183 | 151
Not Completed | 40 | 43 | 72
Not completed — Did not receive study drug | 7 | 12 | 11
Not completed — Adverse Event | 23 | 19 | 37
Not completed — Rejection | 0 | 1 | 16
Not completed — Non-compliance | 4 | 2 | 5
Not completed — Graft Failure | 3 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 4 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Converted to rapamycin | 1 | 0 | 0
Not completed — Acute tubular necrosis | 1 | 0 | 0
Not completed — Incorrect study drug dispensed | 0 | 1 | 0
Not completed — Crossover secondary to possible toxicity | 0 | 1 | 0
Not completed — Poor absorption | 0 | 1 | 0
Not completed — Pancreas transplant | 0 | 0 | 1
Period: Clinical Continuation Phase
Arm/Group | Tacrolimus | Tacrolimus Modified Release | Cyclosporine
Started | 179 | 182 (One participant did not enter the Clinical Continuation phase) | 151
Completed | 9 | 4 | 11
Not Completed | 170 | 178 | 140
Not completed — Adverse Event | 12 | 21 | 14
Not completed — Non-compliance | 8 | 6 | 7
Not completed — Withdrawal by Subject | 22 | 3 | 22
Not completed — Lost to Follow-up | 6 | 3 | 6
Not completed — Graft Failure | 5 | 5 | 2
Not completed — Rejection | 1 | 2 | 2
Not completed — Sponsor discontinued study | 113 | 129 | 79
Not completed — Immunosuppressive treatment crossover | 0 | 3 | 6
Not completed — Physician Decision | 1 | 3 | 0
Not completed — Unable to return to site for study visit | 1 | 0 | 1
Not completed — Pancreas transplant | 1 | 0 | 0
Not completed — Ran out of study drug due to Hurricane | 0 | 1 | 0
Not completed — Discharged to nursing home | 0 | 1 | 0
Not completed — Incorrect study drug dispensed | 0 | 1 | 0
Not completed — Patient opted out | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set; all randomized patients who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tacrolimus | Tacrolimus Modified Release | Cyclosporine | Total
Number analyzed (Participants) | 212 | 214 | 212 | 638
Age Continuous [Mean (Standard Deviation); unit: years] — Demographic data provided for the full analysis set, defined as all randomized patients who received at least one dose of study drug.
  years | 48.62 (12.855) | 47.84 (12.995) | 47.63 (12.953) | 48.03 (12.921)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 76 | 82 | 234
  Male | 136 | 138 | 130 | 404
Race/Ethnicity, Customized [Number; unit: participants]
  White | 152 | 160 | 163 | 475
  Black | 51 | 41 | 36 | 128
  Asian | 5 | 5 | 8 | 18
  Other | 4 | 8 | 5 | 17
Primary Diagnosis [Number; unit: participants]
  Nephrosclerosis/ Hypertensive Nephropathy | 54 | 56 | 43 | 153
  Diabetic Nephropathy | 46 | 38 | 46 | 130
  Glomerulonephritis | 44 | 43 | 43 | 130
  Polycycstic Kidney Disease | 20 | 26 | 20 | 66
  Tubular/ Interstitial Disease | 9 | 5 | 16 | 30
  Systemic Vasculitis | 9 | 10 | 7 | 26
  Congenital/ Hereditary Nephropathy | 7 | 7 | 13 | 27
  Reflux | 1 | 0 | 1 | 2
  Unknown | 17 | 24 | 17 | 58
  Other | 5 | 5 | 6 | 16
Previous Transplant [Number; unit: participants]
  No | 205 | 206 | 203 | 614
  Yes | 7 | 8 | 9 | 24

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Efficacy Failure
Description: Efficacy failure is defined as any participant who died, experienced a graft failure (permanent return to dialysis [> 30 days] or retransplant), had a biopsy-confirmed (Banff Grade ≥ I) acute rejection (BCAR), or was lost to follow-up.
  Biopsies were graded according to the 1997 Banff criteria:
  Borderline: No intimal arteritis present but foci of mild tubulitis; Grade I: Significant interstitial infiltration and foci of moderate to severe tubulitis; Grade II: Mild to severe intimal arteritis Grade III: Transmural arteritis and/or arterial fibrinoid change and necrosis of medial smooth muscle cells with accompanying lymphocytic infiltrate in vessel.
Time Frame: one year
Population: The number of participants analyzed represents the full analysis set, defined as all randomized patients who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus | Tacrolimus Modified Release | Cyclosporine
Number analyzed (Participants) | 212 | 214 | 212
percentage of participants | 15.1 | 14.0 | 17.0
Statistical Analysis 1: Comparison: Tacrolimus vs Cyclosporine; Test type: Non-Inferiority or Equivalence — The non-inferiority margin for this study was pre-specified as 10%; Incidence Difference = -1.9, 95.2% CI 2-sided [-8.9 to 5.2]
Statistical Analysis 2: Comparison: Tacrolimus Modified Release vs Cyclosporine; Test type: Non-Inferiority or Equivalence — The non-inferiority margin for this study was pre-specified as 10%; Incidence Difference = -3.0, 95.2% CI 2-sided [-9.9 to 4.0]

2. Secondary Outcome: Patient Survival at One Year
Description: Patient survival is defined as any participant who is known to be alive one year after the skin closure date. Participants who died or whose outcome was unknown at one year were considered to be non-survivors.
Time Frame: One year
Population: The number of participants analyzed represents the full analysis set.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus | Tacrolimus Modified Release | Cyclosporine
Number analyzed (Participants) | 212 | 214 | 212
percentage of participants | 93.9 | 97.2 | 97.2
Statistical Analysis 1: Comparison: Tacrolimus vs Cyclosporine; Test type: Non-Inferiority or Equivalence — The non-inferiority margin for this study was pre-specified as 10%; Incidence Difference = -3.3, 95% CI 2-sided [-7.2 to 0.6]
Statistical Analysis 2: Comparison: Tacrolimus Modified Release vs Cyclosporine; Test type: Non-Inferiority or Equivalence — The non-inferiority margin for this study was pre-specified as 10%; Incidence Difference = 0.0, 95% CI 2-sided [-3.1 to 3.2]

3. Secondary Outcome: Graft Survival at One Year
Description: Graft survival defined as any participant who did not meet the criteria for graft loss, where graft loss is defined as any re-transplant, permanent return to dialysis (> 30 days), patient death, or participant whose outcome at one year was unknown.
  Participants were only counted once regardless of how many criteria were met.
Time Frame: One year
Population: The number of participants analyzed represents the full analysis set.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus | Tacrolimus Modified Release | Cyclosporine
Number analyzed (Participants) | 212 | 214 | 212
percentage of participants | 91.5 | 95.3 | 95.3
Statistical Analysis 1: Comparison: Tacrolimus vs Cyclosporine; Test type: Non-Inferiority or Equivalence — The non-inferiority margin for this study was pre-specified as 10%; Incidence Difference = -3.8, 95% CI 2-sided [-8.5 to 0.9]
Statistical Analysis 2: Comparison: Tacrolimus Modified Release vs Cyclosporine; Test type: Non-Inferiority or Equivalence — The non-inferiority margin for this study was pre-specified as 10%; Incidence Difference = 0.0, 95% CI 2-sided [-4.0 to 4.1]

4. Secondary Outcome: Percentage of Participants With Biopsy Confirmed Acute Rejection at 6 and 12 Months
Description: Rejection episodes were confirmed by biopsy by the clinical site pathologist. Biopsies were graded according to the 1997 Banff criteria:
  Borderline: No intimal arteritis present but foci of mild tubulitis; Grade I: Significant interstitial infiltration and foci of moderate to severe tubulitis; Grade II: Mild to severe intimal arteritis Grade III: Transmural arteritis and/or arterial fibrinoid change and necrosis of medial smooth muscle cells with accompanying lymphocytic infiltrate in vessel.
  Acute rejection is defined as a grade ≥ I.
Time Frame: Six months and 12 months
Population: The number of participants analyzed represents the full analysis set.
Measure: Number; unit: percentage of participants
Arm/Group | Tacrolimus | Tacrolimus Modified Release | Cyclosporine
Number analyzed (Participants) | 212 | 214 | 212
percentage of participants
  At 6 Months | 3.8 | 7.9 | 11.8
  At 12 Months | 7.5 | 10.3 | 13.7
Statistical Analysis 1: Comparison: Tacrolimus vs Cyclosporine; Comparison of tacrolimus with cyclosporine at 6 months; Test type: Non-Inferiority or Equivalence — The non-inferiority margin for this study was pre-specified as 10%; Incidence Difference at 6 Months = -8.0, 95% CI 2-sided [-13.1 to -3.0]
Statistical Analysis 2: Comparison: Tacrolimus Modified Release vs Cyclosporine; Comparison of Tacrolimus Modified Release with Cyclosporine at 6 months; Test type: Non-Inferiority or Equivalence — The non-inferiority margin for this study was pre-specified as 10%; Incidence Difference at 6 Months = -3.8, 95% CI 2-sided [-9.5 to 1.8]
Statistical Analysis 3: Comparison: Tacrolimus vs Cyclosporine; Comparison of tacrolimus with cyclosporine at 12 months; Test type: Non-Inferiority or Equivalence — The non-inferiority margin for this study was pre-specified as 10%; Incidence Difference at 12 Months = -6.1, 95% CI 2-sided [-12.0 to -0.3]
Statistical Analysis 4: Comparison: Tacrolimus Modified Release vs Cyclosporine; Comparison of Tacrolimus Modified Release with Cyclosporine at 12 months; Test type: Non-Inferiority or Equivalence — The non-inferiority margin for this study was pre-specified as 10%; Incidence Difference at 12 months = -3.4, 95% CI 2-sided [-9.6 to 2.8]

5. Secondary Outcome: Time to First Biopsy-confirmed Acute Rejection Episode
Description: Time to first biopsy-confirmed acute rejection episode defined as the number of days from skin closure (Day 0) to the date of biopsy. Rejection episodes were confirmed by biopsy by the clinical site pathologist and graded according to the 1997 Banff criteria:
  Borderline: No intimal arteritis present but foci of mild tubulitis; Grade I: Significant interstitial infiltration and foci of moderate to severe tubulitis; Grade II: Mild to severe intimal arteritis Grade III: Transmural arteritis and/or arterial fibrinoid change and necrosis of medial smooth muscle cells with accompanying lymphocytic infiltrate in vessel.
  Acute rejection is defined as a grade ≥ I.
Time Frame: one year
Population: The number of participants analyzed represents the full analysis set.
Measure: Median (Full Range); unit: days
Arm/Group | Tacrolimus | Tacrolimus Modified Release | Cyclosporine
Number analyzed (Participants) | 212 | 214 | 212
days | 156.00 [3.0 to 316.0] | 11.00 [6.0 to 327.0] | 52.00 [1.0 to 311.0]

6. Secondary Outcome: Number of Participants Requiring Anti-lymphocyte Antibody Therapy for Treatment of Rejection
Description: Rejection episodes were confirmed by biopsy by the clinical site pathologist. Participants with histologically-proven Banff Grade II or III rejection or participants with steroid-resistant rejection were treated with anti-lymphocyte antibody treatment according to institutional practice.
  Biopsies were graded according to the 1997 Banff criteria:
  Borderline: No intimal arteritis present but foci of mild tubulitis; Grade I: Significant interstitial infiltration and foci of moderate to severe tubulitis; Grade II: Mild to severe intimal arteritis Grade III: Transmural arteritis and/or arterial fibrinoid change and necrosis of medial smooth muscle cells with accompanying lymphocytic infiltrate in vessel.
Time Frame: one year
Population: The number of participants analyzed represents the full analysis set.
Measure: Number; unit: participants
Arm/Group | Tacrolimus | Tacrolimus Modified Release | Cyclosporine
Number analyzed (Participants) | 212 | 214 | 212
participants | 6 | 8 | 18

7. Secondary Outcome: Severity of Acute Rejection
Description: Rejection episodes were confirmed by biopsy by the clinical site pathologist. Biopsies were graded according to the 1997 Banff criteria:
  Borderline: No intimal arteritis present but foci of mild tubulitis; Grade IA: Significant interstitial infiltration and foci of moderate tubulitis; Grade IB: Significant interstitial infiltration and foci of severe tubulitis; Grade IIA: Mild to moderate intimal arteritis in at least 1 arterial cross section Grade IIB: Severe intimal arteritis comprising >25% of the luminal area lost in at least 1 arterial cross section; Grade III: Transmural arteritis and/or arterial fibrinoid change and necrosis of medial smooth muscle cells with accompanying lymphocytic infiltrate in vessel.
Time Frame: one year
Population: The number of participants analyzed represents the full analysis set with a biopsy-confirmed acute rejection episode during one year.
Measure: Number; unit: participants
Arm/Group | Tacrolimus | Tacrolimus Modified Release | Cyclosporine
Number analyzed (Participants) | 16 | 22 | 29
participants
  Grade I-A | 8 | 11 | 14
  Grade I-B | 4 | 3 | 6
  Grade II-A | 3 | 6 | 6
  Grade II-B | 1 | 1 | 1
  Grade III | 0 | 1 | 2

8. Secondary Outcome: Number of Participants Experiencing Multiple Rejection Episodes
Description: This analysis includes rejection episodes that were either confirmed by biopsy by the clinical site pathologist or were clinically treated.
Time Frame: one year
Population: The number of participants analyzed represents the full analysis set.
Measure: Number; unit: participants
Arm/Group | Tacrolimus | Tacrolimus Modified Release | Cyclosporine
Number analyzed (Participants) | 212 | 214 | 212
participants | 2 | 4 | 8

9. Secondary Outcome: Number of Participants With Clinically Treated Acute Rejection Episodes
Description: A clinically treated acute rejection episode was any biopsy-confirmed or suspected rejection episode that was treated with immunosuppressive therapy.
Time Frame: one year
Population: The number of participants analyzed represents the full analysis set.
Measure: Number; unit: participants
Arm/Group | Tacrolimus | Tacrolimus Modified Release | Cyclosporine
Number analyzed (Participants) | 212 | 214 | 212
participants | 25 | 39 | 45

10. Secondary Outcome: Number of Participants With Treatment Failure
Description: Treatment failure was defined as the discontinuation of randomized study drug for any reason. Participants who met the definition of treatment failure were to be followed throughout the 12-month treatment period.
Time Frame: one year
Population: The number of participants analyzed represents the full analysis set.
Measure: Number; unit: participants
Arm/Group | Tacrolimus | Tacrolimus Modified Release | Cyclosporine
Number analyzed (Participants) | 212 | 214 | 212
participants | 33 | 31 | 61

11. Secondary Outcome: Number of Participants Who Crossed Over Due to Treatment Failure
Description: Participants were allowed to cross over to an alternative primary immunosuppressive regimen (either to the tacrolimus or cyclosporine treatment arms) to address an adverse event which led to randomized study drug discontinuation or in the case of severe or refractory rejection. Crossover to the modified release tacrolimus treatment arm was not permitted.
Time Frame: one year
Population: The number of participants analyzed represents the full analysis set.
Measure: Number; unit: participants
Arm/Group | Tacrolimus | Tacrolimus Modified Release | Cyclosporine
Number analyzed (Participants) | 212 | 214 | 212
participants | 6 | 10 | 39

12. Secondary Outcome: Change From Month 1 in Serum Creatinine at Month 6 and Month 12
Description: Renal function was assessed by the change from Month 1 in serum creatinine six months and 12 months after transplant.
Time Frame: Month 1, Month 6, and Month 12
Population: The number of participants analyzed represents the full analysis set with available data at Month 1 and at each time point.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Tacrolimus | Tacrolimus Modified Release | Cyclosporine
Number analyzed (Participants) | 212 | 214 | 212
mg/dL
  At 6 months [N=184, 184, 169] | -0.09 (0.63) | -0.08 (0.56) | -0.01 (0.53)
  At 12 months [N=173, 182, 147] | -0.08 (0.76) | -0.14 (0.62) | -0.04 (0.53)

13. Secondary Outcome: Change From Month 1 in Creatinine Clearance at Month 6 and Month 12
Description: Renal function was assessed by creatinine clearance, calculated using the Cockcroft-Gault formula.
Time Frame: Month 1, Month 6, and Month 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Tacrolimus | Tacrolimus Modified Release | Cyclosporine
Number analyzed (Participants) | 212 | 214 | 212
mL/min
  At 6 months [N=184, 184, 167] | 0.83 (13.77) | 0.47 (12.90) | -1.79 (14.09)
  At 12 months [N=173, 182, 145] | 1.50 (16.07) | 2.62 (14.32) | -0.25 (14.54)

14. Secondary Outcome: Kaplan-Meier Estimate of Patient Survival at the End of the Study
Description: Patient survival was defined as any participant who was alive at the end of the study. Patient survival was censored at the time of last follow-up contact.
Time Frame: End of study (maximum time on study was 1,941 days).
Population: The number of participants analyzed represents the full analysis set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus | Tacrolimus Modified Release | Cyclosporine
Number analyzed (Participants) | 212 | 214 | 212
percentage of participants | 91.2 [86.8 to 95.7] | 93.2 [89.7 to 96.8] | 91.7 [87.7 to 95.8]
Statistical Analysis 1: Comparison: Tacrolimus vs Cyclosporine; Test type: Superiority or Other; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-6.5 to 5.5]
Statistical Analysis 2: Comparison: Tacrolimus Modified Release vs Cyclosporine; Test type: Superiority or Other; Mean Difference (Final Values) = 1.5, 95% CI 2-sided [-3.9 to 6.9]

15. Secondary Outcome: Kaplan-Meier Estimate of Graft Survival at the End of the Study
Description: Graft survival was defined as any participant who did not meet the definition of graft loss, where graft loss was any retransplant or the permanent return to dialysis (more than 30 days) or patient death.
  Graft survival was censored at the time of last follow-up contact.
Time Frame: End of study (maximum time on study was 1,941 days).
Population: The number of participants analyzed represents the full analysis set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus | Tacrolimus Modified Release | Cyclosporine
Number analyzed (Participants) | 212 | 214 | 212
percentage of participants | 82.7 [76.9 to 88.4] | 84.7 [79.0 to 90.4] | 83.9 [78.6 to 89.3]
Statistical Analysis 1: Comparison: Tacrolimus vs Cyclosporine; Test type: Superiority or Other; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-9.1 to 6.6]
Statistical Analysis 2: Comparison: Tacrolimus Modified Release vs Cyclosporine; Test type: Superiority or Other; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [-7.1 to 8.6]

ADVERSE EVENTS:
Time Frame: Up to 1941 days
Arm/Group | Tacrolimus | Tacrolimus Modified Release | Cyclosporine
Serious Adverse Events (participants affected / at risk) | 148/212 | 141/214 | 139/212
Other Adverse Events (participants affected / at risk) | 208/212 | 212/214 | 208/212
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tacrolimus (N=212) | Tacrolimus Modified Release (N=214) | Cyclosporine (N=212)
Cytomegalovirus infection (Infections and infestations) | 15 | 11 | 11
Urinary tract infection (Infections and infestations) | 15 | 11 | 15
Human polyomavirus infection (Infections and infestations) | 9 | 5 | 1
Sepsis (Infections and infestations) | 6 | 8 | 4
Gastroenteritis viral (Infections and infestations) | 5 | 0 | 1
Urosepsis (Infections and infestations) | 5 | 5 | 5
Cellulitis (Infections and infestations) | 4 | 5 | 4
Gastroenteritis (Infections and infestations) | 4 | 14 | 3
Pneumonia (Infections and infestations) | 4 | 10 | 7
Pyelonephritis (Infections and infestations) | 4 | 5 | 3
Bronchitis (Infections and infestations) | 3 | 2 | 1
Escherichia urinary tract infection (Infections and infestations) | 3 | 6 | 5
Herpes zoster (Infections and infestations) | 3 | 3 | 1
Strongyloidiasis (Infections and infestations) | 3 | 0 | 0
Urinary tract infection bacterial (Infections and infestations) | 3 | 3 | 4
Bacteraemia (Infections and infestations) | 2 | 2 | 2
Bacterial pyelonephritis (Infections and infestations) | 2 | 2 | 0
Cytomegalovirus colitis (Infections and infestations) | 2 | 0 | 0
Cytomegalovirus viraemia (Infections and infestations) | 2 | 2 | 0
Endocarditis (Infections and infestations) | 2 | 0 | 0
Osteomyelitis (Infections and infestations) | 2 | 2 | 1
Subcutaneous abscess (Infections and infestations) | 2 | 0 | 0
Urinary tract infection enterococcal (Infections and infestations) | 2 | 1 | 1
Abdominal abscess (Infections and infestations) | 1 | 0 | 0
Abscess (Infections and infestations) | 1 | 0 | 0
Abscess limb (Infections and infestations) | 1 | 0 | 1
Bronchitis acute (Infections and infestations) | 1 | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0 | 0
Catheter related infection (Infections and infestations) | 1 | 0 | 0
Catheter sepsis (Infections and infestations) | 1 | 1 | 0
Clostridial infection (Infections and infestations) | 1 | 0 | 1
Clostridium colitis (Infections and infestations) | 1 | 2 | 1
Diabetic foot infection (Infections and infestations) | 1 | 0 | 2
Diarrhoea infectious (Infections and infestations) | 1 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 1 | 1
Furuncle (Infections and infestations) | 1 | 0 | 1
Infected cyst (Infections and infestations) | 1 | 0 | 0
Infected skin ulcer (Infections and infestations) | 1 | 3 | 0
Klebsiella bacteraemia (Infections and infestations) | 1 | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 1 | 1
Localised infection (Infections and infestations) | 1 | 3 | 1
Lung infection pseudomonal (Infections and infestations) | 1 | 0 | 0
Mastoiditis (Infections and infestations) | 1 | 0 | 0
Mycobacterium avium complex infection (Infections and infestations) | 1 | 0 | 0
Orchitis (Infections and infestations) | 1 | 1 | 1
Otitis media (Infections and infestations) | 1 | 0 | 0
Pharyngotonsillitis (Infections and infestations) | 1 | 0 | 0
Pneumonia fungal (Infections and infestations) | 1 | 0 | 0
Pneumonia staphylococcal (Infections and infestations) | 1 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 2
Skin bacterial infection (Infections and infestations) | 1 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 1 | 0
Streptococcal sepsis (Infections and infestations) | 1 | 0 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0 | 0
Tuberculosis (Infections and infestations) | 1 | 0 | 1
Urinary tract infection fungal (Infections and infestations) | 1 | 0 | 0
Urinary tract infection pseudomonal (Infections and infestations) | 1 | 0 | 0
Vancomycin resistant enterococcal infection (Infections and infestations) | 1 | 0 | 0
Viral infection (Infections and infestations) | 1 | 1 | 1
Vulval abscess (Infections and infestations) | 1 | 0 | 0
Wound infection (Infections and infestations) | 1 | 1 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 0
Cellulitis gangrenous (Infections and infestations) | 0 | 0 | 1
Choriomeningitis lymphocytic (Infections and infestations) | 0 | 1 | 0
Condyloma acuminatum (Infections and infestations) | 0 | 1 | 0
Cytomegalovirus gastritis (Infections and infestations) | 0 | 1 | 2
Cytomegalovirus oesophagitis (Infections and infestations) | 0 | 1 | 0
Endocarditis bacterial (Infections and infestations) | 0 | 0 | 1
Gastritis fungal (Infections and infestations) | 0 | 1 | 0
Groin infection (Infections and infestations) | 0 | 1 | 0
Helicobacter gastritis (Infections and infestations) | 0 | 1 | 0
Herpes virus infection (Infections and infestations) | 0 | 0 | 1
Herpetic gingivostomatitis infection (Infections and infestations) | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 4 | 1
Meningitits aseptic (Infections and infestations) | 0 | 0 | 1
Meningitits cryptococcal (Infections and infestations) | 0 | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 2 | 0
Papilloma viral infection (Infections and infestations) | 0 | 1 | 0
Parvovirus infection (Infections and infestations) | 0 | 1 | 1
Perinephric abscess (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Phlebitis infective (Infections and infestations) | 0 | 1 | 0
Pneumonia haemophilus (Infections and infestations) | 0 | 1 | 0
Pneumonia klebsiella (Infections and infestations) | 0 | 1 | 0
Postoperative abscess (Infections and infestations) | 0 | 1 | 0
Postoperative infection (Infections and infestations) | 0 | 1 | 2
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 | 0 | 1
Streptococcal infection (Infections and infestations) | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1
Urinary tract infection staphylococcal (Infections and infestations) | 0 | 0 | 1
Vaginitis (Infections and infestations) | 0 | 0 | 1
Varicella (Infections and infestations) | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 12 | 10 | 3
Vomiting (Gastrointestinal disorders) | 8 | 8 | 5
Nausea (Gastrointestinal disorders) | 7 | 6 | 3
Abdominal pain (Gastrointestinal disorders) | 5 | 2 | 5
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 2 | 2 | 0
Diverticulitis (Gastrointestinal disorders) | 2 | 3 | 1
Enterocutaneous fistula (Gastrointestinal disorders) | 2 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal wall cyst (Gastrointestinal disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 1
Diarhoea haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 2
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis due to biliary obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Peritoneal haematoma (Gastrointestinal disorders) | 1 | 0 | 0
Rectal polyp (Gastrointestinal disorders) | 1 | 0 | 0
Rectal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Subileus (Gastrointestinal disorders) | 1 | 1 | 1
Umbilical hernia obstructive (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal haematoma (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 | 0 | 3
Abdominal wall disorder (Gastrointestinal disorders) | 0 | 1 | 0
Acute abdomen (Gastrointestinal disorders) | 0 | 1 | 0
Appendicitis perforated (Gastrointestinal disorders) | 0 | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 2
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 2
Gastric ulcer haemorhage (Gastrointestinal disorders) | 0 | 0 | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 1 | 0
Gingival hyperplasia (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 2 | 2
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Oesophageal erosion (Gastrointestinal disorders) | 0 | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1
Peritonitis (Gastrointestinal disorders) | 0 | 2 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 0 | 1
Salivary gland enlargement (Gastrointestinal disorders) | 0 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Complications of transplant surgery (Injury, poisoning and procedural complications) | 5 | 3 | 2
Graft dysfunction (Injury, poisoning and procedural complications) | 5 | 3 | 2
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 5 | 2 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0
Foot Fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 2 | 1 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 1 | 0
Arteriovenous graft site complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cardiac pacemaker malfunction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 1 | 1 | 2
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1 | 1
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Perinephric collection (Injury, poisoning and procedural complications) | 1 | 1 | 2
Perirenal haematoma (Injury, poisoning and procedural complications) | 1 | 1 | 1
Post procedural discharge (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural urine leak (Injury, poisoning and procedural complications) | 1 | 2 | 1
Postoperative haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 1
Renal haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 2 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Burns third degree (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Graft complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Haematuria traumatic (Injury, poisoning and procedural complications) | 0 | 0 | 1
Incision site complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Medical device compilation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pubic rami fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Renal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 2 | 2
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 3 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound secretion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 9 | 10 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 5 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 5 | 5 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 4 | 2 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 6 | 4
Fluid overload (Metabolism and nutrition disorders) | 2 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 2 | 2 | 0
Diabetic foot (Metabolism and nutrition disorders) | 1 | 2 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 4 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1
Diabetes with hyperosmolarity (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 18 | 11 | 15
Blood in stool (Investigations) | 1 | 1 | 0
Blood urea increased (Investigations) | 1 | 0 | 0
Cardiac stress test abnormal (Investigations) | 1 | 0 | 1
Haematocrit decreased (Investigations) | 1 | 0 | 0
Haemaglobin decreased (Investigations) | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0
Volume blood decreased (Investigations) | 1 | 0 | 0
Blood creatine increased (Investigations) | 0 | 1 | 0
Blood glucose increased (Investigations) | 0 | 0 | 1
Cytomegalovirus test positive (Investigations) | 0 | 0 | 1
International normalized ration increased (Investigations) | 0 | 0 | 1
Urine output decreased (Investigations) | 0 | 1 | 3
Weight decreased (Investigations) | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 9 | 4 | 7
Renal Impairment (Renal and urinary disorders) | 4 | 3 | 3
Hydronephrosis (Renal and urinary disorders) | 3 | 2 | 4
Dysuria (Renal and urinary disorders) | 2 | 0 | 2
Haematuria (Renal and urinary disorders) | 2 | 4 | 4
Obstructive uropathy (Renal and urinary disorders) | 2 | 0 | 0
Renal insufficiency (Renal and urinary disorders) | 2 | 5 | 0
Urinary incontinence (Renal and urinary disorders) | 2 | 0 | 0
Bladder disorder (Renal and urinary disorders) | 1 | 0 | 0
Bladder neck obstruction (Renal and urinary disorders) | 1 | 0 | 0
Haemorrhage urinary tract (Renal and urinary disorders) | 1 | 0 | 0
Nephropathy (Renal and urinary disorders) | 1 | 0 | 0
Renal vein thrombosis (Renal and urinary disorders) | 1 | 1 | 1
Ureteric obstruction (Renal and urinary disorders) | 1 | 0 | 1
Ureteric stenosis (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 1 | 2
Acute prerenal failure (Renal and urinary disorders) | 0 | 0 | 1
Azotaemia (Renal and urinary disorders) | 0 | 1 | 0
Hydroureter (Renal and urinary disorders) | 0 | 0 | 1
Nephropathy Toxic (Renal and urinary disorders) | 0 | 0 | 1
Nephrotic Syndrome (Renal and urinary disorders) | 0 | 0 | 1
Pelvi-ureteric obstruction (Renal and urinary disorders) | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1
Renal artery stenosis (Renal and urinary disorders) | 0 | 0 | 1
Renal artery thrombosis (Renal and urinary disorders) | 0 | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 0 | 0 | 1
Stress incontinence (Renal and urinary disorders) | 0 | 1 | 0
Urethral meatus stenosis (Renal and urinary disorders) | 0 | 1 | 0
Urethral obstruction (Renal and urinary disorders) | 0 | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 1
Urinoma (Renal and urinary disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 5 | 4 | 4
Coronary artery disease (Cardiac disorders) | 4 | 0 | 1
Angina pectoris (Cardiac disorders) | 3 | 0 | 1
Cardiac arrest (Cardiac disorders) | 3 | 1 | 2
Cardiac failure congestive (Cardiac disorders) | 3 | 6 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 3 | 3
Cardiac failure (Cardiac disorders) | 2 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0
Aortic valve incompetence (Cardiac disorders) | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 1 | 2 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0
Right ventricular failure (Cardiac disorders) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 1
Angina unstable (Cardiac disorders) | 0 | 1 | 0
Aortic valve disease (Cardiac disorders) | 0 | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 0 | 0 | 1
Atrioventricular block (Cardiac disorders) | 0 | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 1 | 0
Cardio respiratory arrest (Cardiac disorders) | 0 | 2 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Coronary artery insufficiency (Cardiac disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1
Ventricular bigeminy (Cardiac disorders) | 0 | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 7 | 4 | 4
Haematoma (Vascular disorders) | 2 | 1 | 2
Hypotension (Vascular disorders) | 2 | 5 | 2
Lymphocele (Vascular disorders) | 2 | 1 | 4
Arterial thrombosis limb (Vascular disorders) | 1 | 0 | 0
Arterivenous Fistula, acquired (Vascular disorders) | 1 | 0 | 0
Gangrene (Vascular disorders) | 1 | 2 | 2
Lymphorrhoea (Vascular disorders) | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 2 | 1
Peripheral artery dissection (Vascular disorders) | 1 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 1 | 0
Thrombosis (Vascular disorders) | 1 | 2 | 0
Vascular Insufficency (Vascular disorders) | 1 | 0 | 0
Aortic aneurysm (Vascular disorders) | 0 | 2 | 0
Arterial stenosis limb (Vascular disorders) | 0 | 1 | 0
Atherosclerosis (Vascular disorders) | 0 | 2 | 0
Femoral arterial stenosis (Vascular disorders) | 0 | 1 | 0
Femoral artery occlusion (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 3
Hypertensive crisis (Vascular disorders) | 0 | 3 | 2
Iliac artery stenosis (Vascular disorders) | 0 | 0 | 2
Intermittent Claudication (Vascular disorders) | 0 | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 1 | 0
Peripheral artery aneurysm (Vascular disorders) | 0 | 1 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1 | 0
Peripheral occlusive disease (Vascular disorders) | 0 | 1 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 1
Renovascular Hypertension (Vascular disorders) | 0 | 0 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 0 | 1
Venous stenosis (Vascular disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Acute Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chronic Obstructive airways Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chronic Obstructive airways Disease exacerbated (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea exacerbated (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Maxillary sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 6 | 4 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2 | 0
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 3
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Haemolysis (Blood and lymphatic system disorders) | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Pyrexia (General disorders) | 5 | 5 | 8
Chest pain (General disorders) | 2 | 4 | 0
Oedema peripheral (General disorders) | 2 | 1 | 0
Adhesion (General disorders) | 1 | 0 | 0
Asthenia (General disorders) | 1 | 2 | 1
Impaired healing (General disorders) | 1 | 2 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0 | 0
Anasarca (General disorders) | 0 | 2 | 0
Catheter site haemorrhage (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 2 | 0
Oedema (General disorders) | 0 | 1 | 0
Rigors (General disorders) | 0 | 1 | 0
Sudden death (General disorders) | 0 | 1 | 0
Swelling (General disorders) | 0 | 0 | 1
Ulcer haemorrhage (General disorders) | 0 | 1 | 0
Convulsion (Nervous system disorders) | 3 | 1 | 1
Dizziness (Nervous system disorders) | 2 | 0 | 0
Headache (Nervous system disorders) | 2 | 3 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0
Diabetic hypersmolar coma (Nervous system disorders) | 1 | 1 | 0
Dysaesthesia (Nervous system disorders) | 1 | 0 | 0
Guillain Barre syndrome (Nervous system disorders) | 1 | 0 | 0
Sleep apnoea syndrome (Nervous system disorders) | 1 | 0 | 0
Sleep paralysis (Nervous system disorders) | 1 | 0 | 0
Viith nerve paralysis (Nervous system disorders) | 1 | 0 | 0
Cerebellar haemorrhage (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 2
Encephalitis (Nervous system disorders) | 0 | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0
Multiple sclerosis (Nervous system disorders) | 0 | 0 | 1
Neuropathy (Nervous system disorders) | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0
Normal pressure hydrocephalus (Nervous system disorders) | 0 | 1 | 0
Parkinson's disease (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 2
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2 | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Carcinoid tumour of the pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Carcinoid tumour of the appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Carcinoid tumour of the stomach (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lymphooroliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Monoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Bone Spur (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Fracture malunion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc space narrowing (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Localized osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spondylosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 3 | 3 | 0
Mental status changes (Psychiatric disorders) | 2 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Completed Suicide (Psychiatric disorders) | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 2 | 0
Hallucination (Psychiatric disorders) | 0 | 1 | 0
Major depression (Psychiatric disorders) | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0
Epididymitis (Reproductive system and breast disorders) | 1 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0
Scrotal oedema (Reproductive system and breast disorders) | 1 | 1 | 0
Testicular infarction (Reproductive system and breast disorders) | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 1
Gynaecomastia (Reproductive system and breast disorders) | 0 | 1 | 0
Ovarian cyst torsion (Reproductive system and breast disorders) | 0 | 1 | 0
Pelvic muscles inadequate (Reproductive system and breast disorders) | 0 | 1 | 0
Priapism (Reproductive system and breast disorders) | 0 | 1 | 0
Prostatis (Reproductive system and breast disorders) | 0 | 3 | 0
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 | 1 | 0
Knee arthoplasty (Surgical and medical procedures) | 1 | 0 | 0
Nephrectomy (Surgical and medical procedures) | 1 | 1 | 0
Pancreas transplant (Surgical and medical procedures) | 1 | 1 | 1
Parathyroidectomy (Surgical and medical procedures) | 1 | 0 | 0
Umbilical hernia repair (Surgical and medical procedures) | 1 | 1 | 0
Abdominal hernia repair (Surgical and medical procedures) | 0 | 0 | 1
Abdominal panniculectomy (Surgical and medical procedures) | 0 | 1 | 0
Abdominoplasty (Surgical and medical procedures) | 0 | 1 | 0
Cholecystectomy (Surgical and medical procedures) | 0 | 1 | 0
Colostomy closure (Surgical and medical procedures) | 0 | 0 | 1
Coronary arterial stent insertion (Surgical and medical procedures) | 0 | 1 | 0
Hip arthroplasty (Surgical and medical procedures) | 0 | 1 | 0
Hospitalisation (Surgical and medical procedures) | 0 | 0 | 1
Inguinal hernia repair (Surgical and medical procedures) | 0 | 0 | 1
Small intestinal resection (Surgical and medical procedures) | 0 | 0 | 1
Hyperparathyroidism tertiary (Endocrine disorders) | 3 | 1 | 0
Goitre (Endocrine disorders) | 1 | 0 | 0
Hyperparathyroidism (Endocrine disorders) | 1 | 1 | 1
Bile duct stone (Hepatobiliary disorders) | 2 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 2 | 2
Biliary colic (Hepatobiliary disorders) | 0 | 1 | 0
Biliary dilatation (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 3 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic lesion (Hepatobiliary disorders) | 0 | 1 | 0
Graft loss (Immune system disorders) | 1 | 0 | 1
Kidney transplant rejection (Immune system disorders) | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 1 | 0 | 1
Anomalous pulmonary venous connection (Congenital, familial and genetic disorders) | 0 | 1 | 0
Retinitis (Eye disorders) | 1 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Murder (Social circumstances) | 1 | 0 | 0
Treatment noncompliance (Social circumstances) | 0 | 1 | 0
Deafness (Ear and labyrinth disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tacrolimus (N=212) | Tacrolimus Modified Release (N=214) | Cyclosporine (N=212)
Diarrhoea (Gastrointestinal disorders) | 91 | 94 | 53
Constipation (Gastrointestinal disorders) | 68 | 85 | 82
Nausea (Gastrointestinal disorders) | 71 | 74 | 90
Vomiting (Gastrointestinal disorders) | 49 | 51 | 46
Dyspepsia (Gastrointestinal disorders) | 36 | 32 | 32
Abdominal pain (Gastrointestinal disorders) | 22 | 26 | 35
Abdominal pain upper (Gastrointestinal disorders) | 21 | 16 | 18
Flatulence (Gastrointestinal disorders) | 22 | 15 | 14
Abdominal distension (Gastrointestinal disorders) | 15 | 11 | 18
Loose stools (Gastrointestinal disorders) | 14 | 11 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 9 | 12
Haemorrhoids (Gastrointestinal disorders) | 5 | 12 | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 59 | 50 | 45
Hypomagnesaemia (Metabolism and nutrition disorders) | 57 | 52 | 44
Hyperkalaemia (Metabolism and nutrition disorders) | 48 | 40 | 38
Hyperlipidaemia (Metabolism and nutrition disorders) | 35 | 35 | 52
Hyperglycaemia (Metabolism and nutrition disorders) | 37 | 30 | 28
Hypokalaemia (Metabolism and nutrition disorders) | 31 | 31 | 33
Diabetes mellitus (Metabolism and nutrition disorders) | 20 | 25 | 9
Hypocalcaemia (Metabolism and nutrition disorders) | 15 | 13 | 25
Metabolic acidosis (Metabolism and nutrition disorders) | 12 | 15 | 11
Hypercholesterolaemia (Metabolism and nutrition disorders) | 10 | 8 | 16
Fluid overload (Metabolism and nutrition disorders) | 14 | 9 | 9
Dehydration (Metabolism and nutrition disorders) | 16 | 10 | 4
Dyslipidaemia (Metabolism and nutrition disorders) | 4 | 12 | 6
Oedema peripheral (General disorders) | 72 | 75 | 97
Fatigue (General disorders) | 22 | 32 | 26
Oedema (General disorders) | 27 | 17 | 25
Pyrexia (General disorders) | 20 | 21 | 28
Asthenia (General disorders) | 22 | 16 | 22
Chest pain (General disorders) | 16 | 19 | 12
Pain (General disorders) | 8 | 11 | 14
Anasarca (General disorders) | 8 | 12 | 4
Tremor (Nervous system disorders) | 73 | 75 | 42
Headache (Nervous system disorders) | 50 | 45 | 52
Dizziness (Nervous system disorders) | 27 | 21 | 23
Paraesthesia (Nervous system disorders) | 3 | 12 | 13
Hypoaesthesia (Nervous system disorders) | 5 | 8 | 11
Incision site complication (Injury, poisoning and procedural complications) | 46 | 31 | 42
Post procedural pain (Injury, poisoning and procedural complications) | 42 | 27 | 37
Graft dysfunction (Injury, poisoning and procedural complications) | 41 | 27 | 31
Post procedural discharge (Injury, poisoning and procedural complications) | 6 | 10 | 12
Complications of transplant surgery (Injury, poisoning and procedural complications) | 11 | 5 | 10
Anaemia (Blood and lymphatic system disorders) | 59 | 68 | 55
Leukopenia (Blood and lymphatic system disorders) | 33 | 35 | 25
Polycythaemia (Blood and lymphatic system disorders) | 13 | 12 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 27 | 32 | 29
Arthralgia (Musculoskeletal and connective tissue disorders) | 26 | 27 | 28
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 27 | 27 | 26
Muscle Cramp (Musculoskeletal and connective tissue disorders) | 17 | 20 | 22
Osteopenia (Musculoskeletal and connective tissue disorders) | 12 | 13 | 13
Hypertension (Vascular disorders) | 63 | 59 | 69
Hypotension (Vascular disorders) | 17 | 19 | 17
Orthostatic Hypotension (Vascular disorders) | 9 | 15 | 5
Urinary tract infection (Infections and infestations) | 49 | 30 | 42
Upper respiratory tract infection (Infections and infestations) | 24 | 27 | 29
Oral Candidiasis (Infections and infestations) | 9 | 15 | 13
Sinusitis (Infections and infestations) | 7 | 15 | 5
Blood creatinine increased (Investigations) | 41 | 32 | 36
Weight increased (Investigations) | 18 | 14 | 22
Blood magnesium decreased (Investigations) | 19 | 15 | 12
Urine output decreased (Investigations) | 8 | 12 | 10
Blood phosphorus decreased (Investigations) | 10 | 11 | 6
Cardiac Murmur (Investigations) | 11 | 7 | 5
Insomnia (Psychiatric disorders) | 60 | 52 | 45
Anxiety (Psychiatric disorders) | 23 | 27 | 21
Depression (Psychiatric disorders) | 13 | 11 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 | 27 | 26
Cough (Respiratory, thoracic and mediastinal disorders) | 26 | 15 | 21
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 15 | 16 | 11
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 12 | 10 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 20 | 24 | 15
Acne (Skin and subcutaneous tissue disorders) | 13 | 18 | 22
Alopecia (Skin and subcutaneous tissue disorders) | 15 | 14 | 4
Rash (Skin and subcutaneous tissue disorders) | 10 | 11 | 5
Dysuria (Renal and urinary disorders) | 23 | 15 | 20
Haematuria (Renal and urinary disorders) | 18 | 15 | 20
Proteinuria (Renal and urinary disorders) | 5 | 13 | 10
Tachycardia (Cardiac disorders) | 11 | 9 | 10
Hirsutism (Endocrine disorders) | 0 | 0 | 18

LIMITATIONS AND CAVEATS:
Company makes no warranties or representations of any kind as to the posting, expressed or implied, including warranties of merchantability and fitness for a particular purpose, and shall not be liable for any damages.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data or until 18 months have elapsed following study completion. Sponsor must receive a site's manuscript at least 30 days prior to publication to ensure that no confidential information of Sponsor is included in the document.